CLINICAL TRIAL: NCT06758739
Title: Comparison of Curcumin and Intralesional Steroids in Oral Submucous Fibrosis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Hafiza Sara Adrees, Post Graduate Resident OMFS, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U111-1315-4100
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Oral Submucous Fibrosis
Keywords: Potentially Malignant Disorder; Oral Submucous Fibrosis; Intralesional Steroids; Curcumin; Anti-Inflammatory; Anti-Fibrotic
MeSH Terms: conditions — Oral Submucous Fibrosis | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): The Group A will undergo curcumin treatment for oral submucous Fibrosis. In Group A curcumin capsule (500 mg) will be given two per day. Patient will receive 1000 mg curcumin per day and will be assessed month on month basis for three months.
  Interventions: Drug: Curcumin (Turmeric)
- Group B (Experimental): The Group B will undergo Intralesional Steroids treatment in oral submucous fibrosis. In Group B Intralesional Steroid Injection will be administered weekly and assessed on monthly basis for three months.
  Interventions: Drug: Intralesional Steroid Injection

INTERVENTIONS:
Drug: Curcumin (Turmeric) — Curcumin Capsule will be given two per day for three months. Patient Recovery progress will be monitored month on month basis for consecutive three month.
  Arms: Group A
Drug: Intralesional Steroid Injection — Intralesional Steroid Injection (1cc), one per week, will be administered in the fibrous bands wherever formed in the oral cavity. Patient recovery progress will be monitored on monthly basis for three months.
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to learn if Curcumin is better than Intralesional Steroid Injection for the treatment of oral submucous fibrosis. The main question it aims to answers are:

1. If Curcumin is more effective to improve burning sensation as compared to Intralesional steroid.
2. Does Curcumin treatment results in better mouth opening versus Intralesional steroid.
3. Can Curcumin helps to improve tongue protrusion as compared to Intralesional steroids.

Participants will be:

* Assessed for one month, two month and three month.
* Burning Sensation will be assessed with visual analogue scale (VAS).
* Mouth Opening will be measured in mm with ruler.
* Tongue Protrusion will be assessed with the visual analogue scale (VAS).

DETAILED DESCRIPTION:
Objective:

To compare the efficacy of Curcumin versus Intralesional steroids in term of burning sensation, mouth opening and tongue Protrusion

Hypothesis:

Curcumin is more effective in terms of burning sensation, mouth opening (interincisal distance) and tongue Protrusion as compared to intralesional steroids.

Operational Definitions:

Oral submucous fibrosis is chronic, slowly progressive precancerous condition caused by areca nut characterized by restricted mouth opening, burning sensation, stiffness and blanching of mucosa and limitation of tongue Protrusion9. It will be clinically assessed as difficulty in mouth opening, burning sensation, fibrous bands & blanching of mucosa along with limited tongue movement.

Efficacy:

Efficacy of Curcumin & intralesional steroids will be assessed in terms of burning sensation VAS score, mouth opening & Tongue Protrusion

Burning Sensation:

A burning sensation in oral submucous fibrosis is often due to tissue changes, dryness, nutritional deficiencies, or secondary infections affecting the oral mucosa. Patient feels pain or discomfort in mouth especially when eating hot or spicy food Patient will be asked for burning sensation & based on severity numerical score given by VAS (Visual Analog Scale) (Bohra et al.)9

Mouth Opening:

Mouth opening is progressively restricted due to fibroses and stiffness of oral tissue. It will be measured in mm. Patient will be asked to open mouth as wide as he/she can & with the help of mental scale & divider (Vernier caliper) between maxillary incisor & mandibular incisor9.

Tongue Protrusion:

Tongue Protrusion in oral submucous fibrosis refers to the difficulty or inability to fully move the tongue out of the mouth due to stiffness and restricted mobility caused by fibrotic changes in the oral tissues. It will be assessed from normal mesio-incisal angel of maxillary central incisor to the tip of tongue when maximally extended with wide mouth open (Ramesh et al.)11

Material and Methods:

Study Design:

Randomized Central trial (RCT)

Study Setting:

Department of Oral & Maxillofacial surgery, Services Institute of Medical Sciences Lahore

Duration of Study:

Six months

Sample Size: A sample size will be of 70 patients (35 in each group). Calculated using the expected mean difference of burning sensation VAS score between curcumin group and intralesional steroids inj.

Sampling Technique:

Non-probability purposive sampling technique.

Sample Selection:

Inclusion Criteria:

Patients diagnosed with Oral submucous fibrosis in accordance with operational definition.

Male & Female

Exclusion Criteria:

Patient unable to quit the habit of gutkha, tobacco & betel nut chewing Patient With uncontrolled diabetes Patient with chronic kidney disease Pregnant female Patient with untreated malignancy/taking immunosuppressant drugs Patient with H/O ORAL SUBMUCOUS FIBROSIS in last months

Data Collection Procedure:

All eligible patients undergoing oral submucous fibrosis treatment will be invited to participate in the study and informed consent will be obtained from all the volunteer participants. Total 70 (35 in each group) will be randomized into two equal size groups i.e. Group A and B by using online computer-generated program which concealed randomization and treatment allocation. A structured Proforma will be used to call demographic and clinical data. Before treatment, baseline burning sensation, mouth opening (interincisal distance) and tongue Protrusion will be noted. In group A, Patient will receive Curcumin Capsule (nutrifactor) 2 per day for 3 months. In group B, Patient will receive intralesional steroid injection 4mg/1cc weekly for 3 months. Participants health care provider, data collector and outcome assessors will be blinded to the treatment allocation. Patient will be assessed for burning sensation, INTERINCISAL DISTANCE & tongue protrusion monthly. As per operational definitions, efficacy in terms of burning sensation VAS score, greater inter Incisal distance & tongue Protrusion will be compared between Curcumin and Intralesional steroid groups.

Data Collection Tools:

All Study variables will be assessed by single person at Month 1, Month 2 and Month 3 post clinical trial. Clinical parameters will be assessed through proforma designed in English as well as in Local language.

Data Analysis Procedure:

Statistical Package for Social Sciences (SPSS) version 27 will be used for data entry & analysis. The quantitative variables such as age, burning sensation VAS score, mouth opening & tongue Protrusion, will reported using mean ± standard deviation. The quantitative variable such as gender will be reported using percent. The baseline profile between groups will be compared using student t-test. The improvement within the group by the end of 1st, 2nd & 3rd month will be tabulated & analyzed. The clinical improvement of a particular regimen (within the same group) before & after treatment will be analyzed using paired t-test. The improvement observed serially within the same group will be evaluated using repeated measures ANOVA. Comparisons between the two groups will be done using unpaired t-test.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Oral submucous fibrosis in accordance with operational definition.
* Male & Female

Exclusion Criteria:

* Patient unable to quit the habit of gutkha, tobacco & betel nut chewing
* Patient With uncontrolled diabetes
* Patient with chronic kidney disease
* Pregnant female
* Patient with untreated malignancy/taking immunosuppressant drugs
* Patient with H/O ORAL SUBMUCOUS FIBROSIS in last months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Mean of Burning Sensation | Monthl 1, Month 2, Month 3
  A burning sensation in oral submucous fibrosis is often due to tissue changes, dryness, nutritional deficiencies, or secondary infections affecting the oral mucosa. Patient will be asked for burning sensation & based on severity numerical score given by VAS (Visual Analog Scale) 0-100.
Mean of Mouth Opening | Month 1, Month 2, Month 3
  Mouth opening is progressively restricted due to fibroses and stiffness of oral tissue. It will be measured in mm. Patient will be asked to open mouth as wide as he/she can & with the help of metal scale & divider (Vernier caliper) between maxillary incisor & mandibular incisor.
Mean of Tongue Protrusion | Month 1, Month 2, Month 3
  Tongue Protrusion in oral submucous fibrosis refers to the difficulty or inability to fully move the tongue out of the mouth. It will be assessed from normal mesio-incisal angel of maxillary central incisor to the tip of tongue when maximally extended with wide mouth open by Visual Analogue Scale (VAS) 0-100.

CONTACTS AND LOCATIONS:
Locations (1):
- Services Institute of Medical Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kerr AR, Warnakulasuriya S, Mighell AJ, Dietrich T, Nasser M, Rimal J, Jalil A, Bornstein MM, Nagao T, Fortune F, Hazarey VH, Reichart PA, Silverman S, Johnson NW. A systematic review of medical interventions for oral submucous fibrosis and future research opportunities. Oral Dis. 2011 Apr;17 Suppl 1:42-57. doi: 10.1111/j.1601-0825.2011.01791.x. PMID 21382138
- [Background] Roques C, Teot L. The use of corticosteroids to treat keloids: a review. Int J Low Extrem Wounds. 2008 Sep;7(3):137-45. doi: 10.1177/1534734608320786. Epub 2008 Jul 8. PMID 18611924
- [Background] Ramesh, D.N.S.V., Saba N. lycopene and combination of lycopene with multivitamins in the treatment of oral submucous fibrosis patients - A comparative study. Int. J Curr Res. 2017;9:53177-82.
- [Background] Piyush P, Mahajan A, Singh K, Ghosh S, Gupta S. Comparison of therapeutic response of lycopene and curcumin in oral submucous fibrosis: A randomized controlled trial. Oral Dis. 2019 Jan;25(1):73-79. doi: 10.1111/odi.12947. Epub 2018 Aug 22. PMID 30059188
- [Background] Bohra A, Maheswari TNU, Harsh A, Garg A. Black Turmeric and Aloe Vera in the Management of Oral Submucous Fibrosis: A Prospective Clinical Study. Asian Pac J Cancer Prev. 2021 Dec 1;22(12):3941-3947. doi: 10.31557/APJCP.2021.22.12.3941. PMID 34967575
- [Background] Yadav M, Aravinda K, Saxena VS, Srinivas K, Ratnakar P, Gupta J, Sachdev AS, Shivhare P. Comparison of curcumin with intralesional steroid injections in Oral Submucous Fibrosis - A randomized, open-label interventional study. J Oral Biol Craniofac Res. 2014 Sep-Dec;4(3):169-73. doi: 10.1016/j.jobcr.2014.11.003. Epub 2014 Nov 20. PMID 25737939
- [Background] Nagpal M, Sood S. Role of curcumin in systemic and oral health: An overview. J Nat Sci Biol Med. 2013 Jan;4(1):3-7. doi: 10.4103/0976-9668.107253. PMID 23633828
- [Background] Zhang SS, Gong ZJ, Li WH, Wang X, Ling TY. Antifibrotic effect of curcumin in TGF-beta 1-induced myofibroblasts from human oral mucosa. Asian Pac J Cancer Prev. 2012;13(1):289-94. doi: 10.7314/apjcp.2012.13.1.289. PMID 22502687
- [Background] Aziz SR. Coming to America: betel nut and oral submucous fibrosis. J Am Dent Assoc. 2010 Apr;141(4):423-8. doi: 10.14219/jada.archive.2010.0194. PMID 20354091
- [Background] Nigam NK, Aravinda K, Dhillon M, Gupta S, Reddy S, Srinivas Raju M. Prevalence of oral submucous fibrosis among habitual gutkha and areca nut chewers in Moradabad district. J Oral Biol Craniofac Res. 2014 Jan-Apr;4(1):8-13. doi: 10.1016/j.jobcr.2013.10.005. Epub 2013 Nov 20. PMID 25737912
- [Background] Rajendran R, Deepthi K, Nooh N, Anil S. alpha4beta1 integrin-dependent cell sorting dictates T-cell recruitment in oral submucous fibrosis. J Oral Maxillofac Pathol. 2011 Sep;15(3):272-7. doi: 10.4103/0973-029X.86678. PMID 22144828
- [Background] Pindborg JJ, Sirsat SM. Oral submucous fibrosis. Oral Surg Oral Med Oral Pathol. 1966 Dec;22(6):764-79. doi: 10.1016/0030-4220(66)90367-7. No abstract available. PMID 5224185
- [Background] Hazarey VK, Erlewad DM, Mundhe KA, Ughade SN. Oral submucous fibrosis: study of 1000 cases from central India. J Oral Pathol Med. 2007 Jan;36(1):12-7. doi: 10.1111/j.1600-0714.2006.00485.x. PMID 17181736